CLINICAL TRIAL: NCT04071509
Title: Pilot Study on the Prevention of PNX (Pneumothorax) and Haemorrhagic Complications in Diagnostic Percutaneous Lung Biopsy Procedures Using the MIPP-Kit Device.
Brief Title: Prevention of PNX and Haemorrhagic Complications in Diagnostic Percutaneous Lung Biopsy Using the MIPP-Kit Device
Acronym: MIPP-PNX1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BetaGlue Technologies spa (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MIPP-PNX1
Record Dates: First submitted 2018-05-19; First posted 2019-08-28 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2019-08

CONDITIONS: Complications in Diagnostic Percutaneous Lung Biopsy Procedures
Keywords: Lung Biopsy, pneumothorax, interventional radiology
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percutaneous Lung Biopsy (Experimental)
  Interventions: Device: Percutaneous Lung Biopsy

INTERVENTIONS:
Device: Percutaneous Lung Biopsy — Patients will undergo the usual biopsy procedure with a fine needle inserted through a larger guide needle, under CT guidance; at the end of the biopsy, the MIPP-Kit will be introduced through the same guide needle. The guide needle and the MIPP Kit will be retracted together slowly, whilst injecting BioGlue in appropriate amounts along the whole track, from the lesion to the skin.

SUMMARY:
The study will assess the safety and feasibility of a new medical device, MIPP-Kit, for the prevention of complications during diagnostic, CT guided ,percutaneous lung needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for diagnostic percutaneous lung biopsy

Exclusion Criteria:

* Pregnant, or breastfeeding patient (Female)
* actively participating in other clinical trials in the previous 30 days
* known allergies to the investigational device components
* comorbidities that preclude undergoing percutaneous lung biopsy procedure
* concomitant treatments that preclude undergoing percutaneous lung biopsy procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-27 (Actual)

PRIMARY OUTCOMES:
Rate of complications associated with percutaneous lung biopsy | 48 hours after procedure
  incidence of clinical complications commonly associated with lung biopsy (pneumothorax and haemorrhage)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Istituto Tumori Bari Giovanni Paolo II, Bari
  - Fondazione Policlinico Universitario A. Gemelli, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gadaleta CD, Iezzi R, Tanzilli A, Puppini G, Carriero PL, Amato A. Pilot clinical study on the prevention of complications after lung biopsy by the MIPP kit PNX device. Transl Cancer Res. 2022 Dec;11(12):4338-4348. doi: 10.21037/tcr-22-1203. PMID 36644169